CLINICAL TRIAL: NCT01313442
Title: Acquisition of Data, Blood, and Tumor Tissue Samples From Patients With Gastrointestinal Cancer
Brief Title: Acquisition of Blood and Tumor Tissue Samples From Patients With Gastrointestinal Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110112; 11-C-0112
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2026-01-12 (Actual); Status verified 2025-10-07

CONDITIONS: Non-GI Cancers; Cancer of Gastrointestinal Tract; Gastrointestinal Cancer
Keywords: Gut Microbiota; Analysis of immune subsets with regard to their function; Samples; Natural History; Gastrointestinal Cancer; Gastrointestinal Tract Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/ Cohort 1: Individuals with a diagnosis of cancer

SUMMARY:
Background:

- Gastrointestinal cancers can occur in the throat, stomach, gallbladder, liver, pancreas, and colon. Researchers are interested in evaluating how active the immune system is in trying to fight the cancer by studying blood and tumor tissue donated from individuals who have been diagnosed with gastrointestinal cancers.

Objectives:

- To collect blood and tumor samples from individuals who have been diagnosed with gastrointestinal cancers in order to study the immune system s response to the cancer.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with throat, stomach, gallbladder, liver, pancreatic, or colon cancer, and are scheduled to be treated at the National Institutes of Health.

Design:

* The study will require at least one but no more than four visits to the National Institutes of Health Clinical Center.
* Participants will be screened with a physical examination and medical history, and will provide a baseline blood sample for study.
* Participants will provide additional blood samples 2 and 4 months after the baseline sample, as well as a final sample at the completion of the treatment protocol.
* Participants will provide tumor tissue samples only if they undergo a surgical procedure related to the treatment for their gastrointestinal cancer.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
BACKGROUND:

* Numerous recent therapeutic advances have changed standard treatment options for patients with GI cancer. These include newer chemotherapeutic agents in addition to established proof of principle for anti-angiogenic agents. The burden of GI cancers is reflected by the presence of three GI cancer types in the top five causes of cancer mortality. Over 58,000 deaths yearly can be attributed to GI cancer.
* While immune-based therapies in GI cancers are experimental at the current time, a gathering body of literature is suggestive of an enormous potential, either alone, or most likely in combination with standard chemotherapy.
* Before immunotherapy can be combined with non-immune based treatment options we first need to investigate the effects of non-immune based therapies on immune responses (especially immune-evasive mechanisms) with cancer.
* Commensal gut microbiota play an important role in colonic inflammation and colon cancer. The human gut flora consists of approximately 100 trillion microbial cells, which their disruption leads to many types of diseases including inflammatory bowel disease and colorectal cancer. Recent studies have shown that colon cancer patients as well other patients with gastrointestinal cancers have an altered gut flora when compared to healthy controls. As an example, intestinal microbiome has been shown to contribute to the start and progression of certain kinds of liver diseases such as NAFLD as well as end-stage liver diseases 2-4 Therefore, it is important to investigate further as to how the gut affects the patient's response to chemotherapy, other types of cancer therapy and to tumor growth in general.

OBJECTIVES:

To serve as an umbrella protocol to allow collection, storage and investigation of samples from patients with gastrointestinal (GI) cancers in support of Thoracic and GI Oncology Branch translational trials to develop new therapeutic agents and novel treatment approaches as well as new prognostic and diagnostic models. Also, to collect samples from patients with non-GI cancers for comparison.

ELIGIBILITY:

* Individuals undergoing evaluation for participation in NCI treatment protocols in the NCI intramural program with diagnosis of cancer.
* 18 year of age or older.

DESIGN:

* Blood, tumor tissue or stool samples may be collected from consenting participants at the initial visit and/or at the time of visit to NIH, scheduled per other NIH protocols.
* Analysis of participant's samples include but not limited to immune-monitoring, single cell sequencing, identifying of gene expression and generation of CAR-T cells.
* Stool samples will be used to determine the intestinal microbiome.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Individuals 18 years of age and older
* Individuals with a diagnosis of cancer
* Individuals must be able to understand and willing to sign a written informed consent document

EXCLUSION CRITERIA:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2011-03-02 (Actual)

PRIMARY OUTCOMES:
Collected samples | 10 years
  Collected blood, tumor samples from participants with gastrointestinal (GI) cancers being reviewed by Medical Oncology Branch and to perform immune studies

CONTACTS AND LOCATIONS:
Overall Officials: Tim F Greten, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.@@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Greten TF, Ormandy LA, Fikuart A, Hochst B, Henschen S, Horning M, Manns MP, Korangy F. Low-dose cyclophosphamide treatment impairs regulatory T cells and unmasks AFP-specific CD4+ T-cell responses in patients with advanced HCC. J Immunother. 2010 Feb-Mar;33(2):211-8. doi: 10.1097/CJI.0b013e3181bb499f. PMID 20139774
- [Background] Goldszmid RS, Trinchieri G. The price of immunity. Nat Immunol. 2012 Oct;13(10):932-8. doi: 10.1038/ni.2422. Epub 2012 Sep 18. PMID 22990891
- [Background] Iida N, Dzutsev A, Stewart CA, Smith L, Bouladoux N, Weingarten RA, Molina DA, Salcedo R, Back T, Cramer S, Dai RM, Kiu H, Cardone M, Naik S, Patri AK, Wang E, Marincola FM, Frank KM, Belkaid Y, Trinchieri G, Goldszmid RS. Commensal bacteria control cancer response to therapy by modulating the tumor microenvironment. Science. 2013 Nov 22;342(6161):967-70. doi: 10.1126/science.1240527. PMID 24264989
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-C-0112.html